CLINICAL TRIAL: NCT00998751
Title: Phase 2 Study of Oral AB1010 in Non Pre-treated, Inoperable Patients With Locally Advanced/Metastatic Gastro-intestinal Stromal Tumour (GIST)
Brief Title: Masitinib in Locally Advanced/Metastatic Gastro-intestinal Stromal Tumour (GIST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB04016
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Gastro-intestinal Stromal Tumours
Keywords: cKIT inhibitor; GIST
MeSH Terms: interventions — masitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- masitinib (AB1010) (Experimental): oral masitinib 7.5 mg/kg/day
  Interventions: Drug: oral masitinib

INTERVENTIONS:
Drug: oral masitinib — 7.5 mg/kg/day
  Other Names: AB1010

SUMMARY:
The objective is to evaluate the efficacy and safety of AB1010 at 7.5 mg/kg/day in the treatment of non pre-treated, inoperable patients with locally advanced/metastatic GIST.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients, age >18
* Life expectancy > 6 months
* Histological proven, metastatic, or locally advanced and non-operable, non- pre-treated GIST.
* Patients having never received any tyrosine kinase inhibitor, including as adjuvant therapy
* C-Kit (CD117) positive tumors detected immuno-histochemically
* Measurable tumor lesions with longest diameter >20 mm using conventional techniques or >10 mm with spiral CT scan

Exclusion Criteria:

* Documented allergy to the similar drug of AB1010
* Inadequate organ function
* Patients with a history of any other malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate according to Response Evaluation Criteria In Solid Tumors (RECIST) | 2 months

SECONDARY OUTCOMES:
Progression Free Survival | until disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Lecesne, Villejuif, France

REFERENCES:
- [Result] Le Cesne A, Blay JY, Bui BN, Bouche O, Adenis A, Domont J, Cioffi A, Ray-Coquard I, Lassau N, Bonvalot S, Moussy A, Kinet JP, Hermine O. Phase II study of oral masitinib mesilate in imatinib-naive patients with locally advanced or metastatic gastro-intestinal stromal tumour (GIST). Eur J Cancer. 2010 May;46(8):1344-51. doi: 10.1016/j.ejca.2010.02.014. Epub 2010 Mar 6. PMID 20211560